CLINICAL TRIAL: NCT06201533
Title: Effects of Low-intensity Exercise on Cognitive Function, Blood Biomarkers, and Metabolomic Alterations of Older Adults at Risk of Developing Dementia
Brief Title: Low-intensity Physical-cognitive Exercise and Cognitive Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Somporn Sungkarat, Associate Professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RSA660640
Record Dates: First submitted 2023-12-30; First posted 2024-01-11 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Mild Cognitive Impairment
Keywords: mild cognitive impairment; low intensity exercise; cognitive function; fibroblast growth factor 21
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-intensity, combined physical-cognitive exercise (Experimental): The exercise program will be prescribed at low intensity for 50 minutes/session, 3 times /week for 12 consecutive weeks.
  Interventions: Behavioral: combined physical-cognitive exercise
- Control (No Intervention): Participants will be asked to maintain their routine lifestyle throughout the study period.

INTERVENTIONS:
Behavioral: combined physical-cognitive exercise — A combined physical-cognitive exercise will be delivered in the form of exergame, where the participants move their body to interact with the game.
  Arms: Low-intensity, combined physical-cognitive exercise

SUMMARY:
This study aims to examine the effects of low-intensity, combined physical-cognitive exercise on cognitive function of older people with mild cognitive impairment (MCI) and identify the mechanisms by which this exercise protocol exerts cognitive function. Older adults with MCI will be recruited to either an exercise or a control group. Low-intensity, combined physical-cognitive exercise will be prescribed to the exercise group 3 times per week for 3 months while the control group will maintain their routine lifestyle. It is hypothesized that at the end of the trial, participants in the exercise group will demonstrate significant improvement in cognitive performance and circulating biomarkers compared to baseline and the control group.

DETAILED DESCRIPTION:
Accumulating evidence suggests that dementia may be preventable, especially at an early stage. Mild cognitive impairment (MCI), a preclinical phase of dementia, is a potentially reversible condition as several individuals with MCI could revert to normal level of cognition. Exercise has shown promising evidence of neurocognitive protection, however, not all studies reported such benefits. Type and intensity of exercise are two main factors that have often been accounted for discrepancies in previous findings. Based on previous evidence, low-intensity and combined physical-cognitive exercise might give the best result for cognitive enhancement.

Thus, this study aims to examine the effects of low-intensity, combined physical-cognitive training on cognitive function of older people with MCI and identify the mechanisms by which this exercise protocol exerts cognitive function in individuals with MCI. A single-blinded, randomized controlled trial will be conducted. Older adults with MCI will be recruited to either an exercise or a control group. Low-intensity, combined physical-cognitive exercise will be prescribed to the exercise group 3 times per week for 3 months while the control group will maintain their routine lifestyle. Outcome measures will be assessed at baseline and after a 3-month exercise. The primary outcome measures will be cognitive performance (specific and global cognitive function) and plasma brain-derived neurotrophic factor (BDNF). The secondary outcomes will include physical performance (functional mobility and strength), interleukin 6 (IL-6), fibroblast growth factor 21 (FGF21), and metabolomic profiles. Intention-to-treat method will be applied for data analyses.

ELIGIBILITY:
Inclusion Criteria:

* meeting the criteria for MCI (or mNCD) based on the recent DSM-V criteria
* comprehend instructions and able to comply with the study procedures
* not taking any medications for their cognition and not planning to start medications during the study trial

Exclusion Criteria:

* presence of medical condition(s) unsafe to exercise or affect cognition and mobility
* presence of depressive symptoms
* exercise regularly

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-04-07 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
ADAS-Cog | 12 weeks
  Alzheimer's Disease Assessment-cognitive subscale (ADAS-Cog) will be assessed at baseline and 12 weeks. The total scores range from 0-70 with higher scores indicating greater cognitive impairment.
Memory | 12 weeks
  Logical memory test will be evaluated at baseline and 12 weeks.
Executive function | 12 weeks
  Trail making test (TMT) part B-A will be evaluated at baseline and 12 weeks.
Plasma BDNF | 12 weekss
  Level of plasma brain-derived neurotrophic factor will be assessed at baseline and 12 weeks.

SECONDARY OUTCOMES:
Attention | 12 weeks
  Digit span forward-backward will be evaluated at baseline and 12 weeks
Plasma IL-6 | 12 weeks
  Level of plasma IL-6 will be assessed at baseline and 12 weeks.
FGF21 | 12 weeks
  Level of plasma fibroblast growth factor 21 (FGF21) will be assessed at baseline and 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: S Sungkarat, PhD, Principal Investigator — Chiang Mai University
Locations (1):
- Department of Physical Therapy, Faculty of Associated Medical Sciences, Chiang Mai University, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kumfu S, Sungkarat S, Boripantakul S, Sa-Nguanmoo P, Chattipakorn SC. Effects of home-based, low-intensity exergaming on cognitive function of individuals with mild cognitive impairment: a study protocol for a randomized controlled trial. BMC Geriatr. 2025 Jun 4;25(1):408. doi: 10.1186/s12877-025-06054-w. PMID 40468210